CLINICAL TRIAL: NCT00722800
Title: A Single-Center, Randomized Double-Blind, Parallel-Group Study to Examine the Safety and Efficacy of YAZ Compared With Placebo In The Treatment Of Hidradenitis Suppurativa
Brief Title: A Study to Examine the Safety and Efficacy of Drospirenone and Ethinyl Estradiol (YAZ) Versus Placebo In HS
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Poor recruitment
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Bayer (Industry)
Responsible Party: Principal Investigator, Alexandra Kimball, Principal Investigator, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 20080p-000843
Record Dates: First submitted 2008-07-24; First posted 2008-07-28 (Estimated); Results first posted 2014-01-16 (Estimated); Last update posted 2014-02-10 (Estimated); Status verified 2014-01

CONDITIONS: Hidradenitis Suppurativa
Keywords: YAZ; oral contraceptive; hidradenitis suppurativa
MeSH Terms: conditions — Hidradenitis Suppurativa | interventions — drospirenone; Ethinyl Estradiol; drospirenone and ethinyl estradiol combination

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Experimental): drospirenone and ethinyl estradiol
  Interventions: Drug: drospirenone and ethinyl estradiol (YAZ)
- B (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: drospirenone and ethinyl estradiol (YAZ) — 1 tablet daily for 24 weeks
  Arms: A
Drug: Placebo — 1 tablet daily for 24 weeks
  Arms: B

SUMMARY:
The purpose of this study is to find out if taking a birth control pill, YAZ, is safe and effective for treating hidradenitis suppurativa. Hidradenitis suppurativa (HS) is a chronic (long lasting) skin disorder that mostly affects the armpits and groin area. It appears as blackheads and one or more red, tender bumps that may enlarge, break open, and drain pus. Scarring may result after several attacks of the disease.

The exact cause of HS isn't known. However, it is believed that the plugging of hair follicles and bacterial infection that occur in acne also occur in HS. Many of the medications used for treating acne are also used for HS. However, none of the medications are consistently effective.

YAZ is a combination birth control pill. Nearly all birth control pills are made up of a combination of estrogen and progestin hormones. YAZ contains ethinyl estradiol (an estrogen) and drospirenone (a progestin). People who develop acne have sebaceous glands that are over-stimulated by male sex hormones (androgens). Sebaceous glands secrete an oily substance into a hair follicle to lubricate hair or skin. The progestin in YAZ actually blocks the male sex hormones (androgens) that cause acne. Hormones seem to play a role in HS as the condition occurs after puberty. It affects more women than men and HS often gets worse around the time a women has her menstrual period.

YAZ has been approved by the U.S. Food and Drug Administration (FDA) to treat moderate acne in women who desire an oral contraceptive for birth control.

This study uses a placebo. A placebo looks like the study drug but contains no active drug. We use placebos in research studies to learn if the effects seen in research subjects are truly from the study drug or from other reasons.

DETAILED DESCRIPTION:
Hidradenitis suppurativa is a chronic suppurative and scarring disease primarily affecting the axillae and inguinal and perineal areas. The apocrine glands are the primary targets. It is characterized by firm, tender red nodules that soon become fluctuant and painful. Rupture of the lesion, suppuration, formation of sinus tracts and scarring may occur.

The exact etiology of HS remains obscure. Proposed etiologic factors include follicular occlusion and bacterial infection, genetics, host defense defects, hormones, cigarette smoking, and irritants. Hormones seem to play a role, as the condition occurs after puberty, affects more women than men, and often flares in the perimenstrual period.

Treating hidradenitis remains a challenge. Although many patients benefit from long-term treatment with systemic antibiotics (eg, tetracycline, minocycline, clindamycin, erythromycin in combination with metronidazole), no published evidence suggests that the long-term use of antibiotics alters the natural course of HS. Oral isotretinoin has been used, but is effective only in some cases. Some patients have had a beneficial response to biological agents, especially anti-TNF alpha biologicals such as infliximab. Oral contraceptives containing norgestrel or cyproterone acetate, alone or in combination with supplemental cyproterone acetate, spironolactone or dexamethasone (to block adrenal androgen production), have been shown to reduce the frequency and severity of attacks in women.

YAZ is an oral contraceptive that is FDA approved for acne vulgaris. Unlike other progestins, drospirenone has unique antimineralocorticoid (mild diuretic effect) and antiandrogenic properties. The antiandrogenic property of drospirenone means that it blocks the male sex hormones that can cause acne. It is hoped that that YAZ will offer patients with hidradenitis suppurativa a safe and effective therapeutic option.

Subjects will be assigned to a treatment group upon randomization. Bayer HealthCare Pharmaceuticals personnel, investigators, subjects and study nurse/coordinators will be blinded to the study product treatment assignment. The study duration will be 24 weeks with visits at screening, baseline (week 0), week 6, week 12, week 18, and week 24. Lesion counts (total, inflammatory, non-inflammatory) and an ISGA, and photography will be performed on every visit. A physical examination will be done at baseline and Week 24. Safety will be assessed from reported adverse events (AEs).

ELIGIBILITY:
INCLUSION CRITERIA

1. Female Subjects 14-45 years of age who have achieved spontaneous menarche.
2. Clinical diagnosis of hidradenitis suppurativa of stage II or greater on the Hurley scale.
3. Willing and able to understand and sign informed consent.
4. Able to complete study and comply with study procedures.

EXCLUSION CRITERIA

1. Change is use of oral or topical antibiotics in past 90 days.
2. Use of intralesional steroids within 30 days.
3. Use of isotretinoin in past six months.
4. Use of biologics such as Infliximab (Remicade®) or Etanercept (Enbrel®) within the past 3 months or 5 half lives (whichever is shorter).
5. History of renal insufficiency
6. History of hepatic dysfunction
7. History of adrenal Insufficiency
8. History of vascular or metabolic disease including existing or previous arterial thromboembolic diseases (myocardial infarction, stroke), existing or previous venous thromboembolic diseases (deep vein thrombosis, pulmonary embolism), and any condition which could increase the risk to suffer any of the above mentioned disorders
9. History of hypertension
10. History of Diabetes mellitus with vascular involvement
11. Migraine headaches with focal neurological symptoms
12. Major surgery with prolonged immobilization
13. Known or suspected carcinoma of the breast
14. History of Carcinoma of the endometrium or other known or suspected estrogen-dependent neoplasia
15. Undiagnosed abnormal genital bleeding
16. Cholestatic jaundice of pregnancy or jaundice with prior pill use
17. History of Liver tumor (benign or malignant) or active liver disease
18. Smokers
19. Regular intake of medications that may increase potassium levels such as NSAIDS, potassium sparing diuretics, potassium supplementation, ACE inhibitors, Angiotensin-II receptor antagonists, heparin and aldosterone antagonists.
20. Hypersensitivity to any component of the study drug
21. Clinically significant abnormal findings or conditions (other than acne), which might, in the opinion of the Principal Investigator, interfere with study evaluations or pose a risk to subject safety during the study.
22. Subjects who are known to be pregnant or planning a pregnancy.

Ages: 14 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 4 (Actual)
Dates: Start 2008-10; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alexandra B Kimball, MD, MPH, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Clinical Unit for Research Trials in Skin, Boston, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment methods used were Craig's list, Metro and our hospitals email. All subjects were seen at MGH.
Pre-assignment Details: One subject was ineligible because she was taking ibuprofen regularly.
Groups:
- Drospirenone and Ethinyl Estradiol (YAZ): drospirenone and ethinyl estradiol (YAZ) once a day for 6 months
- Placebo Tablets: Placebo tablet once a day for 6 months
Period: Overall Study
Arm/Group | Drospirenone and Ethinyl Estradiol (YAZ) | Placebo Tablets
Started | 2 | 2
Completed | 0 | 2
Not Completed | 2 | 0
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Physician Decision | 1 | 0

BASELINE CHARACTERISTICS:
Population: One subject was excluded because she was regularly taking ibuprofen. The other subject changed her mind about study participation.
Groups:
- Total: Total of all reporting groups
Arm/Group | Drospirenone and Ethinyl Estradiol (YAZ) | Placebo Tablets | Total
Number analyzed (Participants) | 2 | 2 | 4
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 2 | 2 | 4
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 34 (12.73) | 35.5 (14.85) | 34.75 (11.33)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 4
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 2 | 2 | 4

OUTCOME MEASURES:

1. Primary Outcome: Mean Improvement in the Sartorius Severity Score at Month 6.
Description: The Sartorius Severity score reflects changes in hidradenitis suppurative symptoms, namely the number of lesions (abscesses, nodules, and fistulas) and the longest distance between lesions. A total score is derived based on assessments at up to 8 distinct anatomical regions and ranges from 5 to indefinite. Smaller numbers are better scores and indicate less lesion involvement, thus decreases (negative changes) from baseline indicate improvement in severity of disease.
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Drospirenone and Ethinyl Estradiol (YAZ) | Placebo Tablets
Number analyzed (Participants) | 2 | 2
units on a scale | -3.5 (2.1213) | 12 (33.9411)

2. Secondary Outcome: Change From Baseline in VAS Pain Scale at Month 6.
Description: For this pain assessment, the participant indicated the level of average pain experienced over the past 24 hours on a horizontal line, 10 cm in length. A score of 0 indicated "no pain" and a score of 10 indicated "worst pain". The value indicates the change from the baseline participant assessment on the 0 to 10 scale. A negative value indicates a reduction in pain intensity.
Time Frame: 6 months from Baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Drospirenone and Ethinyl Estradiol (YAZ) | Placebo Tablets
Number analyzed (Participants) | 2 | 2
units on a scale | -2.25 (1.06066) | 2 (8.485281)

3. Secondary Outcome: Change From Baseline in Dermatology Life Quality Index (DLQI) Score at Month 6.
Description: Dermatology Life Quality Index (DLQI) Score is a participant-reported outcome consisting of a set of 10 questions regarding the degree to which the participant's skin has affected certain behaviors and quality of life over the last week. Responses to each are: very much, a lot, a little, or not at all. The DLQI score ranges from 0 (best) to 30 (worst).
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: points
Arm/Group | Drospirenone and Ethinyl Estradiol (YAZ) | Placebo Tablets
Number analyzed (Participants) | 2 | 2
points | 3 (1.4142) | 8.5 (19.0919)

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Drospirenone and Ethinyl Estradiol (YAZ) | Placebo Tablets
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/2
Other Adverse Events (participants affected / at risk) | 1/2 | 1/2
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Drospirenone and Ethinyl Estradiol (YAZ) (N=2) | Placebo Tablets (N=2)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Upper respiratory infection (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
fistula with bacterial infection R-axilla (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
Very small sample size.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No